CLINICAL TRIAL: NCT04156308
Title: Effectiveness of the Osteopathic Treatment in Patients With Nonspecific Cervical Pain: Randomized Controlled Pragmatic Clinical Trial
Brief Title: Effectiveness of the Osteopathic Treatment in Patients With Nonspecific Cervical Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Escola D'osteopatia De Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR407/18
Record Dates: First submitted 2019-09-16; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-09

CONDITIONS: Manual Therapies; Neck Pain
Keywords: osteopathy, osteopathic treatment, non-specific
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: A pragmatic experimental comparative trial with three branches of study (osteopathic treatment with 2 different dosages versus active muscle exercise) is proposed.
Who Masked: Participant, Outcomes Assessor
Masking Description: A double masking is proposed. Three active interventions are compared. The patients will be blinded in relation to the study group they belong to, ensuring the masking of the participants.
  The data that is intended to be obtained for its analysis are of a self-reported nature and will be collected and administered by an external investigator not linked to the interventions, ensuring the masking of the evaluator.
  Due to the nature of the interventions, masking of therapists is not possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined exercises+OMT weekly (Experimental): * This group will conduct a home-based pattern of combined exercises based on stretching, active anti-resisted exercises and joint mobility exercises focused on the cervico-dorsal and scapulo-thoracic regions. Whose clinical effectiveness has shown significant positive changes in pain levels and cervical functionality
  * This group will also receive Osteopathic Manipulative Treatment (OMT): exactly 3 sessions with a weekly frequency (with + -2 days of margin: between 5 and 9 days).
  Interventions: Other: Osteopathic Manipulative Treatment (OMT) - Temp1; Other: Combined Exercises
- Combined exercises+OMT once every 3 weeks (Experimental): * This group will conduct a home-based pattern of combined exercises based on stretching, active anti-resisted exercises and joint mobility exercises focused on the cervico-dorsal and scapulo-thoracic regions. Whose clinical effectiveness has shown significant positive changes in pain levels and cervical functionality
  * This group will also receive Osteopathic Manipulative Treatment (OMT): exactly 3 sessions at the rate of one session every 3 weeks (with + -2 days of margin: between 19-23 days).
  Interventions: Other: Osteopathic Manipulative Treatment (OMT) - Temp1; Other: Combined Exercises
- Combined exercises (Experimental): This group will conduct a home-based pattern of combined exercises based on stretching, active anti-resisted exercises and joint mobility exercises focused on the cervico-dorsal and scapulo-thoracic regions. Whose clinical effectiveness has shown significant positive changes in pain levels and cervical functionality.
  Interventions: Other: Combined Exercises

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment (OMT) - Temp1 — A total of 3 techniques selected from a list of 7 available techniques common to all centers will be applied in each session. The choice of techniques will be based on the results of the examination performed, the particularities of the patient and the clinical experience of the osteopath. In each session the techniques can change under the criteria of the osteopath. However, they will always be 3 and always within the list of available techniques.
  Arms: Combined exercises+OMT once every 3 weeks; Combined exercises+OMT weekly
Other: Combined Exercises — A home-based pattern of combined exercises based on stretching, active anti-resisted exercises and joint mobility exercises focused on the cervico-dorsal and scapulo-thoracic regions. Whose clinical effectiveness has shown significant positive changes in pain levels and cervical functionality

SUMMARY:
In Spain cervical pain affects practically 20% of the population annually, while globally it is estimated that between 22% and 77% of the population will suffer cervical pain at some point in their life. Prevalence increases with age, and is more common in women than in men (1.6: 1). Although the natural evolution of cervical pain tends to improve, the rates of recurrence and chronicity are high. And therefore it becomes an anatomical region of interest in relation to the assessment of the effectiveness and / or effectiveness of the osteopathic therapeutic approach. Different studies prove the efficacy of various manual therapy techniques applied on the cervical and / or upper dorsal region, suggesting significant positive changes in cervical pain and mobility levels in patients with nonspecific cervical pain. It is necessary to bear in mind that the reality of the osteopathic approach to the patient is not limited to the use of a single technique, but that the treatment is formed from a set of them. The ultimate goal is to restore mobility and functionality to a specific region, especially taking into account the concepts of individuality and holism.

A pragmatic experimental comparative trial with three branches of study (osteopathic treatment with 2 different dosages versus active muscle exercise) is proposed.

DETAILED DESCRIPTION:
At the beginning of the 1st session, a battery of questions will be made as an anamnesis with the objective of evidencing possible risk factors at the therapeutic level. The presence of one or more risk factors will suppose the exclusion of the patient from the study.

Next, a brief osteopathic musculoskeletal evaluation will be made to the patient. This exploration will follow a standardized protocol for all patients in the experimental groups (1 and 2).

The tests to be carried out will be:

* Observation (standing patient):

  * Assessment of the anterior projection of the head
  * Assessment of the variation in the physiological curves of the spine
* Active test of the cervical spine with the patient in a sitting position.

  o Flexo-Extension / Rotations / Lateral inclinations
* Segmental test of joint mobility of the cervical and dorsal spine (patient in sitting and supine position)
* Passive mobility test of the cervical spine (patient in the supine position):

  * Flexo-Extension / Rotations / Lateral inclinations

The combination of exercises scheduled at home for all groups is based on the conclusions of different studies, and will consist of:

* Self-resisted active exercise in flexion, rotations and inclinations of the cervical spine.
* Active mobility in its maximum travel (without forcing pain) in flexion, rotations and inclinations of the cervical spine.
* Stretching upper trapezius muscles and scalenes.
* Active mobility in circumferential joints of the glenohumeral joint, and in flexo-extension of the thoracic spine.

The work schedule will be carried out for 7 weeks, at a rate of 5 sessions per week.

It will be the patient himself who will keep a diary record of the activity carried out during the weeks that the trial lasts. The diary will be facilitated by the therapists, and in it the exercises to be performed will be indicated.

For groups 1 and 2, a total of 3 techniques selected from a list of 7 available techniques common to all centers will be applied in each session. The choice of techniques will be based on the results of the examination performed, the particularities of the patient and the clinical experience of the osteopath. In each session the techniques can change under the criteria of the osteopath. However, they will always be 3 and always within the list of available techniques.

For groups 1 and 2, a total of 3 techniques selected from a list of 7 available techniques common to all centers will be applied in each session. The choice of techniques will be based on the results of the examination performed, the particularities of the patient and the clinical experience of the osteopath. In each session the techniques can change under the criteria of the osteopath. However, they will always be 3 and always within the list of available techniques.

For groups 1 and 2, a total of 3 techniques selected from a list of 7 available techniques common to all centers will be applied in each session. The choice of techniques will be based on the results of the examination performed, the particularities of the patient and the clinical experience of the osteopath. In each session the techniques can change under the criteria of the osteopath. However, they will always be 3 and always within the list of available techniques.

The OMT (Osteopathic Manipulative Treatment) techniques that may be applied will be the following:

1. Technique of Inhibition of the suboccipital muscles
2. Functional technique for the middle and deep cervical fascia
3. High-speed cervical spine technique (Cervical wheel C1-C6)
4. High-speed technique in the cervico-dorsal junction (prone position)
5. High speed technique in dorsal column (D1-D12) - (Dog Technique)
6. Muscle stretching technique of the diaphragm (supine decubitus)
7. Thorax joint mobility technique (long lever)

Main Variable:

o Neck Disability Index (NDI). The investigators establish the minimum change to be detected (minimum clinically relevant change) at 5 points. The Spanish version of the NDI will be used, validated by Andrade Ortega et al.24

Secondary Variable:

o Degree of general quality of life, through the "SF-36" Health Survey25.

The data will be reported in the form of a report by the patient himself, who will receive via e-mail (whenever possible) or in printed form the questionnaire to be completed and will deliver to the same center in which the intervention has been carried out.

ELIGIBILITY:
Inclusion Criteria:

* The sample will be formed by patients between the ages of 18 and 75 years, who present cervical pain of any intensity and duration, and with a minimum score of 10 points on the Neck Disability Index (NDI)14,15.

Exclusion Criteria:

* Patients who present at the time of recruitment other pathologies or elements that may condition cervical pain, such as: acute shoulder tendinopathy, cervical radiculopathy, chronic diseases of general musculoskeletal involvement (Chronic Fatigue Syndrome and / or Fibromyalgia). Similarly, patients suffering from any type of vertiginous syndrome, who have suffered a whiplash in the last year or who are or have been under treatment for cervical pain in the last 3 months will also be excluded.

The taking of anti-inflammatories by the patient is not taken as a measure of exclusion. If the patient is under pharmacological treatment, it will be recorded and will be taken into account as a co-intervention. However, this treatment will not be modified under any circumstances nor will it be grounds for exclusion from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of osteopathic treatment | 12 weeks
  The effectiveness of osteopathic treatment will be assessed using two health questionnaires ("SF-36" and "NDI") compared to an exercise plan in patients with nonspecific cervical pain.

SECONDARY OUTCOMES:
Temporal Frequency | 12 weeks
  The result of the treatment applied in different temporal frequencies will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Hernandez Amigo, Principal Investigator — Escola Osteopatia de Barcelona
Locations (3):
- Spain (3):
  - IntegroSalus, Cabrils, Barcelona
  - AXIS, Sant Sadurní d'Anoia, Barcelona
  - Clinica Osteopatia Horta, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross A, Langevin P, Burnie SJ, Bedard-Brochu MS, Empey B, Dugas E, Faber-Dobrescu M, Andres C, Graham N, Goldsmith CH, Bronfort G, Hoving JL, LeBlanc F. Manipulation and mobilisation for neck pain contrasted against an inactive control or another active treatment. Cochrane Database Syst Rev. 2015 Sep 23;2015(9):CD004249. doi: 10.1002/14651858.CD004249.pub4. PMID 26397370
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Franke et al. Franke H, Franke J-D, Fryer G. "Osteopathic manipulative treatment for chronic nonspecific neck pain: A systematic review and meta-analysis". International Journal of Osteopathic Medicine. 2015 Dec;18(4):255-67. [doi:10.1186/1471-2474-15-286]
- [Background] Fredin K, Loras H. Manual therapy, exercise therapy or combined treatment in the management of adult neck pain - A systematic review and meta-analysis. Musculoskelet Sci Pract. 2017 Oct;31:62-71. doi: 10.1016/j.msksp.2017.07.005. Epub 2017 Jul 21. PMID 28750310
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Akhter S, Khan M, Ali SS, Soomro RR. Role of manual therapy with exercise regime versus exercise regime alone in the management of non-specific chronic neck pain. Pak J Pharm Sci. 2014 Nov;27(6 Suppl):2125-8. PMID 25410083
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] Sprafka S, Ward RC, Neff D. What characterizes an osteopathic principle? Selected responses to an open question. J Am Osteopath Assoc. 1981 Sep;81(1):29-33. No abstract available. PMID 6895077
- [Background] Pickar JG. Efectos neurofisiológicos de la manipulación vertebral. Osteopatía científica. 2011;6(1):2-18
- [Background] Gonzalez-Alvarez FJ, Valenza MC, Torres-Sanchez I, Cabrera-Martos I, Rodriguez-Torres J, Castellote-Caballero Y. Effects of diaphragm stretching on posterior chain muscle kinematics and rib cage and abdominal excursion: a randomized controlled trial. Braz J Phys Ther. 2016 Jun 16;20(5):405-411. doi: 10.1590/bjpt-rbf.2014.0169. PMID 27333481
- [Background] Andrade Ortega JA, Delgado Martinez AD, Almecija Ruiz R. Validation of the Spanish version of the Neck Disability Index. Spine (Phila Pa 1976). 2010 Feb 15;35(4):E114-8. doi: 10.1097/BRS.0b013e3181afea5d. PMID 20110848
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Result] Palacios-Cena D, Alonso-Blanco C, Hernandez-Barrera V, Carrasco-Garrido P, Jimenez-Garcia R, Fernandez-de-las-Penas C. Prevalence of neck and low back pain in community-dwelling adults in Spain: an updated population-based national study (2009/10-2011/12). Eur Spine J. 2015 Mar;24(3):482-92. doi: 10.1007/s00586-014-3567-5. Epub 2014 Sep 11. PMID 25208501
- [Result] Cote P, Cassidy DJ, Carroll LJ, Kristman V. The annual incidence and course of neck pain in the general population: a population-based cohort study. Pain. 2004 Dec;112(3):267-273. doi: 10.1016/j.pain.2004.09.004. PMID 15561381
- [Result] Casanova-Mendez A, Oliva-Pascual-Vaca A, Rodriguez-Blanco C, Heredia-Rizo AM, Gogorza-Arroitaonandia K, Almazan-Campos G. Comparative short-term effects of two thoracic spinal manipulation techniques in subjects with chronic mechanical neck pain: a randomized controlled trial. Man Ther. 2014 Aug;19(4):331-7. doi: 10.1016/j.math.2014.03.002. Epub 2014 Mar 14. PMID 24679838
- [Result] Salom-Moreno J, Ortega-Santiago R, Cleland JA, Palacios-Cena M, Truyols-Dominguez S, Fernandez-de-las-Penas C. Immediate changes in neck pain intensity and widespread pressure pain sensitivity in patients with bilateral chronic mechanical neck pain: a randomized controlled trial of thoracic thrust manipulation vs non-thrust mobilization. J Manipulative Physiol Ther. 2014 Jun;37(5):312-9. doi: 10.1016/j.jmpt.2014.03.003. Epub 2014 May 28. PMID 24880778
- [Result] Saavedra-Hernandez M, Arroyo-Morales M, Cantarero-Villanueva I, Fernandez-Lao C, Castro-Sanchez AM, Puentedura EJ, Fernandez-de-las-Penas C. Short-term effects of spinal thrust joint manipulation in patients with chronic neck pain: a randomized clinical trial. Clin Rehabil. 2013 Jun;27(6):504-12. doi: 10.1177/0269215512464501. Epub 2012 Nov 5. PMID 23129812
- [Result] Masaracchio M, Cleland JA, Hellman M, Hagins M. Short-term combined effects of thoracic spine thrust manipulation and cervical spine nonthrust manipulation in individuals with mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2013 Mar;43(3):118-27. doi: 10.2519/jospt.2013.4221. Epub 2012 Dec 7. PMID 23221367
- [Result] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Result] Puntumetakul R, Suvarnnato T, Werasirirat P, Uthaikhup S, Yamauchi J, Boucaut R. Acute effects of single and multiple level thoracic manipulations on chronic mechanical neck pain: a randomized controlled trial. Neuropsychiatr Dis Treat. 2015 Jan 12;11:137-44. doi: 10.2147/NDT.S69579. eCollection 2015. PMID 25624764
- [Result] Gross AR, Paquin JP, Dupont G, Blanchette S, Lalonde P, Cristie T, Graham N, Kay TM, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Santaguida PL, Yee AJ, Radisic GG, Hoving JL, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders: A Cochrane review update. Man Ther. 2016 Aug;24:25-45. doi: 10.1016/j.math.2016.04.005. Epub 2016 Apr 20. PMID 27317503

DOCUMENTS (2):
  • Informed Consent Form (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT04156308/ICF_000.pdf
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04156308/Prot_001.pdf